CLINICAL TRIAL: NCT03640819
Title: Pre-ATNEC - A Multicentre Prospective Feasibility Study of Carbon Dye Tattooing of Biopsied Axillary Node and Surgical Localisation in Breast Cancer Patients
Brief Title: Carbon Dye Tattooing of Biopsied Axillary Node in Breast Cancer
Acronym: pre-ATNEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Amit Goyal, Associate Professor, University Hospitals of Derby and Burton NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 241379
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Sentinel Lymph Node; Breast Cancer; Tattoo; Pigmentation; Axilla; Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tattooing of biopsied node (Experimental): The biopsied node will be tattooed at the time of needle biopsy (fine needle aspiration or core biopsy) or separate visit under ultrasound guidance.
  Interventions: Procedure: Tattooing of biopsied node

INTERVENTIONS:
Procedure: Tattooing of biopsied node — Tattooing (marking) of biopsied node with carbon dye (SPOT dye) at the time of fine needle aspiration or core biopsy or separate visit under ultrasound guidance. The dye will be injected in the cortex of the node and the perinodal tissue under ultrasound guidance. Patients will undergo standard (routine) armpit surgery and may receive neoadjuvant chemotherapy as planned by the clinical team. This could be removal of a few lymph glands (sentinel node biopsy) or removal of all the lymph glands (axillary lymph node dissection) in the armpit. The surgeon will try to identify and remove the tattooed lymph gland at the time of planned armpit surgery.
  Other Names: carbon dye (SPOT dye)

SUMMARY:
The primary aim of this prospective, multicentre study is to determine whether the involved node can be marked using black carbon dye and successfully identified at the time of surgery. The secondary aims are to determine the concordance between the tattooed node and sentinel node, migration of black dye into other nodes, and false-negative rate of tattooed node (in patients undergoing ALND after NACT).

DETAILED DESCRIPTION:
Pretreatment evaluation of axillary lymph nodes and marking of biopsied nodes in patients with newly diagnosed breast cancer is becoming routine practice. Tagging of biopsied axillary lymph nodes with metal markers, similar to what is done for suspicious breast lesions, is being adopted in clinical practice. The need to mark a positive axillary lymph node becomes especially relevant in cases where neoadjuvant chemotherapy (NACT) is anticipated so that these nodes may be identified at the time of surgery. Measures that improve both the accuracy of nodal evaluation after NACT and the ability to assess treatment response are desirable in order to tailor therapies for breast cancer treatment. The investigators sought to test tattooing of biopsied axillary lymph nodes with a sterile black carbon suspension (Spot dye). The concept is based on the experience in the gastrointestinal tract wherein tattooing is widely used for marking lesions or tumours biopsied during endoscopy. India ink tattoos of colonic lesions remain identifiable over a long period of time. Spot is routinely used in the UK for tattooing gastrointestinal tract lesions and is used to mark the axillary lymph nodes in breast cancer by some centres in the US and Europe. The intraoperative success of identifying tattooed axillary lymph nodes and their concordance to sentinel nodes will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Male or female
* Patients scheduled to undergo routine fine needle aspiration (FNA) or core biopsy of abnormal axillary lymph node
* Invasive breast cancer
* Written informed consent for the study

Exclusion Criteria:

* Not undergoing surgery or unfit for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Identification rate of tattooed node | 12 months
  Proportion of patients in whom tattooed node/s were identified.

SECONDARY OUTCOMES:
Concordance of tattooed node and sentinel node | 12 months
  Concordance rate: defined as the percent of patients in whomthe tattooed node is the sentinel node.
Migration of black dye into other nodes | 12 months
  The number of black nodes at the time of sentinel node biopsy or axillary lymph node dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goyal, MS, MD, FRCS, Principal Investigator — Royal Derby Hospital, Derby, UK
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom

REFERENCES:
- [Result] Goyal A, Puri S, Marshall A, Valassiadou K, Hoosein MM, Carmichael AR, Erdelyi G, Sharma N, Dunn J, York J. A multicentre prospective feasibility study of carbon dye tattooing of biopsied axillary node and surgical localisation in breast cancer patients. Breast Cancer Res Treat. 2021 Jan;185(2):433-440. doi: 10.1007/s10549-020-05961-3. Epub 2020 Oct 6. PMID 33025481
- [Derived] Ditsch N, Rubio IT, Gasparri ML, de Boniface J, Kuehn T. Breast and axillary surgery in malignant breast disease: a review focused on literature of 2018 and 2019. Curr Opin Obstet Gynecol. 2020 Feb;32(1):91-99. doi: 10.1097/GCO.0000000000000593. PMID 31833973